CLINICAL TRIAL: NCT04353206
Title: A Feasibility Study Assessing the Safety of Multiple Doses of Anti-SARS-CoV-2 Plasma in Mechanically Ventilated Intubated Patients With Respiratory Failure Due to COVID-19
Brief Title: Convalescent Plasma in ICU Patients With COVID-19-induced Respiratory Failure
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The initiation of the expanded access program for convalescent plasma.
Sponsor: Noah Merin (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor-Investigator, Noah Merin, Assistant Professor, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Acute Care CP Consortium Trial
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Covid-19; Sars-CoV2
Keywords: convalescent plasma; Anti-Sars-COV-2 plasma
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intubated COVID-19 patients in the ICU (Experimental): Mechanically ventilated intubated patients with respiratory failure due to COVID-19
  Interventions: Biological: Multiple Doses of Anti-SARS-CoV-2 convalescent plasma

INTERVENTIONS:
Biological: Multiple Doses of Anti-SARS-CoV-2 convalescent plasma — Subjects to receive single or double plasma units infused on day 0 and potentially days 3 and 6.
  Other Names: convalescent plasma; covid-19 convalescent plasma; anti-SARS-CoV-2 convalescent plasma

SUMMARY:
This study will assess the feasibility of administering multiple doses of convalescent plasma (from people who have recovered form SARS-CoV-2) to Covid-19 positive patients in the Intensive Care Unit receiving mechanical ventilation. Donor plasma will not be obtained under this protocol, but all plasma used will follow FDA guidelines for Investigational COVID-19 Convalescent Plasma use.

Patients may receive single or double plasma units infused on days 0, 3, and 6. This decision may be based on availability of blood plasma. The primary objective of this study is feasibility. Feasibility will be assessed based on the proportion of subjects who consent and receive at least one dose of convalescent plasma. The study will be declared 'feasible' if at least 80% of subjects who consent receive at least one dose.

The secondary study endpoint is overall survival at day 60 after first dose of convalescent plasma. Respiratory status and overall clinical status will be reviewed during follow up on days 14, 28, and 60.

DETAILED DESCRIPTION:
Convalescent plasma is an antibody-rich product made from blood donated by people who have recovered from the disease caused by the virus. Prior experience with respiratory viruses and limited data that have emerged from China suggest that convalescent plasma has the potential to lessen the severity or shorten the length of illness caused by COVID-19. It is important that we evaluate this potential therapy in the context of clinical trials.

As such, this study will assess the feasibility of administering multiple doses of convalescent plasma (from people who have recovered form SARS-CoV-2) to Covid-19 positive patients in the Intensive Care Unit receiving mechanical ventilation. Donor plasma will not be obtained under this protocol, but all plasma used will follow FDA guidelines for Investigational COVID-19 Convalescent Plasma use.

This study will be opened across three separate site: Cedars-Sinai Medical Center, Johns Hopkins University, and University of Pittsburgh Medical Center. 30 patients will be recruited at each site. Each site has received its own FDA IND and IRB approval. As such, the following people are serving as sponsor-investigators at their respective institutions.

David Hager, MD PhD, Johns Hopkins University

Noah Merin, MD PhD, Cedars-Sinai Medical Center

Patients may receive single or double plasma units infused on days 0, 3, and 6. This decision may be based on availability of blood plasma. The primary objective of this study is feasibility. Feasibility will be assessed based on the proportion of subjects who consent and receive at least one dose of convalescent plasma. The study will be declared 'feasible' if at least 80% of subjects who consent receive at least one dose.

The secondary study endpoint is overall survival at day 60 after first dose of convalescent plasma. Respiratory status and overall clinical status will be reviewed during follow up on days 14, 28, and 60.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Respiratory failure requiring mechanical ventilation due to COVID-19 induced pneumonia with confirmation via SARS-CoV-2 RT-PCR testing
* PaO2/FiO2 ratio < 300 (or SpO2/FiO2 < 315)
* Bilateral pulmonary infiltrates

Exclusion Criteria:

* Contraindication to transfusion (severe volume overload, history of anaphylaxis to blood products).
* In the opinion of the site investigator or primary clinical care team, anticipated to die within 48 hours.
* Acute or chronic disease/illness that, in the opinion of the site investigator, has an expected life expectancy of less than 28 days unrelated to COVID-19 induced pneumonia (e.g.; stage IV malignancy, neurodegenerative disease, anoxic brain injury, etc.)
* Use of home oxygen at baseline
* Use of home mechanical ventilation at baseline (CPAP or BIPAP without need for oxygen is NOT an exclusion)
* Respiratory failure caused by illness other than SARS-CoV-2
* Other documented uncontrolled infection.
* More than 72 hours have elapsed since first meeting inclusion criteria
* Severe DIC, TTP, or antithrombin III deficiency needing factor replacement, FFP, cryoprecipitate.
* Patient is on Warfarin and it is deemed necessary to maintain therapeutic INR (because the CP will reverse the warfarin effect).
* On dialysis at the time enrollment is considered.
* Active intracranial bleeding.
* Clinically significant myocardial ischemia.
* Prisoner or Incarceration
* Pregnancy or active breast feeding
* Has already received convalescent plasma for COVID-19 infection during current admission
* Current participation in another interventional research study
* Inability or unwillingness of subject or legal surrogate/representative to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-06-27 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who consent to the study and receive at least one dose of convalescent plasma. | 60 days
  Feasibility of administering convalescent plasma to patients in the ICU who are intubated and mechanically ventilated due to COVID-19-induced respiratory failure will be assessed based on the proportion of subjects who consent and receive at least one dose of CP. The study will be declared 'feasible' if at least 80% of subjects who consent receive at least one dose.

SECONDARY OUTCOMES:
Overall survival of patients in the ICU receiving at least once dose of convalescent plasma for Covid-19-induced respiratory failure. | 60 days
  Overall survival (days, until Day 60). This will be quantified as number of trial patients alive at Day 60 after first dose of CP / total number of patients who received at least one dose of CP.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Merin, MD PhD, Principal Investigator — Cedars-Sinai Medical Center; David Hager, MD PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - 8700 Beverly Blvd., Los Angeles, California
  - Johns Hopkins University, Baltimore, Maryland

REFERENCES:
- [Background] Casadevall A, Scharff MD. Return to the past: the case for antibody-based therapies in infectious diseases. Clin Infect Dis. 1995 Jul;21(1):150-61. doi: 10.1093/clinids/21.1.150. PMID 7578724
- [Background] Casadevall A, Dadachova E, Pirofski LA. Passive antibody therapy for infectious diseases. Nat Rev Microbiol. 2004 Sep;2(9):695-703. doi: 10.1038/nrmicro974. PMID 15372080
- [Background] Zhang JS, Chen JT, Liu YX, Zhang ZS, Gao H, Liu Y, Wang X, Ning Y, Liu YF, Gao Q, Xu JG, Qin C, Dong XP, Yin WD. A serological survey on neutralizing antibody titer of SARS convalescent sera. J Med Virol. 2005 Oct;77(2):147-50. doi: 10.1002/jmv.20431. PMID 16121363
- [Background] Sahr F, Ansumana R, Massaquoi TA, Idriss BR, Sesay FR, Lamin JM, Baker S, Nicol S, Conton B, Johnson W, Abiri OT, Kargbo O, Kamara P, Goba A, Russell JB, Gevao SM. Evaluation of convalescent whole blood for treating Ebola Virus Disease in Freetown, Sierra Leone. J Infect. 2017 Mar;74(3):302-309. doi: 10.1016/j.jinf.2016.11.009. Epub 2016 Nov 17. PMID 27867062
- [Background] Casadevall A, Pirofski LA. Antibody-mediated regulation of cellular immunity and the inflammatory response. Trends Immunol. 2003 Sep;24(9):474-8. doi: 10.1016/s1471-4906(03)00228-x. No abstract available. PMID 12967670
- [Background] Casadevall A, Scharff MD. Serum therapy revisited: animal models of infection and development of passive antibody therapy. Antimicrob Agents Chemother. 1994 Aug;38(8):1695-702. doi: 10.1128/AAC.38.8.1695. No abstract available. PMID 7985997
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] Yeh KM, Chiueh TS, Siu LK, Lin JC, Chan PK, Peng MY, Wan HL, Chen JH, Hu BS, Perng CL, Lu JJ, Chang FY. Experience of using convalescent plasma for severe acute respiratory syndrome among healthcare workers in a Taiwan hospital. J Antimicrob Chemother. 2005 Nov;56(5):919-22. doi: 10.1093/jac/dki346. Epub 2005 Sep 23. PMID 16183666
- [Background] Ko JH, Seok H, Cho SY, Ha YE, Baek JY, Kim SH, Kim YJ, Park JK, Chung CR, Kang ES, Cho D, Muller MA, Drosten C, Kang CI, Chung DR, Song JH, Peck KR. Challenges of convalescent plasma infusion therapy in Middle East respiratory coronavirus infection: a single centre experience. Antivir Ther. 2018;23(7):617-622. doi: 10.3851/IMP3243. Epub 2018 Jun 20. PMID 29923831
- [Background] Arabi YM, Hajeer AH, Luke T, Raviprakash K, Balkhy H, Johani S, Al-Dawood A, Al-Qahtani S, Al-Omari A, Al-Hameed F, Hayden FG, Fowler R, Bouchama A, Shindo N, Al-Khairy K, Carson G, Taha Y, Sadat M, Alahmadi M. Feasibility of Using Convalescent Plasma Immunotherapy for MERS-CoV Infection, Saudi Arabia. Emerg Infect Dis. 2016 Sep;22(9):1554-61. doi: 10.3201/eid2209.151164. PMID 27532807
- [Background] van Erp EA, Luytjes W, Ferwerda G, van Kasteren PB. Fc-Mediated Antibody Effector Functions During Respiratory Syncytial Virus Infection and Disease. Front Immunol. 2019 Mar 22;10:548. doi: 10.3389/fimmu.2019.00548. eCollection 2019. PMID 30967872
- [Background] Wan Y, Shang J, Sun S, Tai W, Chen J, Geng Q, He L, Chen Y, Wu J, Shi Z, Zhou Y, Du L, Li F. Molecular Mechanism for Antibody-Dependent Enhancement of Coronavirus Entry. J Virol. 2020 Feb 14;94(5):e02015-19. doi: 10.1128/JVI.02015-19. Print 2020 Feb 14. PMID 31826992
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Background] Crowe JE Jr, Firestone CY, Murphy BR. Passively acquired antibodies suppress humoral but not cell-mediated immunity in mice immunized with live attenuated respiratory syncytial virus vaccines. J Immunol. 2001 Oct 1;167(7):3910-8. doi: 10.4049/jimmunol.167.7.3910. PMID 11564809
- [Background] Guo L, Ren L, Yang S, Xiao M, Chang D, Yang F, Dela Cruz CS, Wang Y, Wu C, Xiao Y, Zhang L, Han L, Dang S, Xu Y, Yang QW, Xu SY, Zhu HD, Xu YC, Jin Q, Sharma L, Wang L, Wang J. Profiling Early Humoral Response to Diagnose Novel Coronavirus Disease (COVID-19). Clin Infect Dis. 2020 Jul 28;71(15):778-785. doi: 10.1093/cid/ciaa310. PMID 32198501
- [Background] Zhao J, Yuan Q, Wang H, Liu W, Liao X, Su Y, Wang X, Yuan J, Li T, Li J, Qian S, Hong C, Wang F, Liu Y, Wang Z, He Q, Li Z, He B, Zhang T, Fu Y, Ge S, Liu L, Zhang J, Xia N, Zhang Z. Antibody Responses to SARS-CoV-2 in Patients With Novel Coronavirus Disease 2019. Clin Infect Dis. 2020 Nov 19;71(16):2027-2034. doi: 10.1093/cid/ciaa344. PMID 32221519
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428